CLINICAL TRIAL: NCT00431886
Title: Usefulness of 64 Slice Multi-Detector Computed Tomography as a First Diagnostic Approach in Acute Chest Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B-0603/031-009
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2007-02

CONDITIONS: Chest Pains
Keywords: Chest pains; Computed tomography; Emergency
MeSH Terms: conditions — Chest Pain; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: 64 multi-detector computed tomography

SUMMARY:
The purpose of this study is to determine the usefulness of 64 slice multi-detector computed tomography as a first diagnostic approach in acute chest pain patients in emergency room

DETAILED DESCRIPTION:
We prospectively enrolled the patients with acute chest pain who visited ED. Exclusion criteria were myocardial infarction (MI) with ST elevation, unstable vital sign, uncontrolled arrhythmia, renal dysfunction, hypersensitivity to contrast media and pregnancy. Patients were allocated into 3 categories based on history, physical exam, and electrocardiogram: 1) definite angina with uncertainty of regarding MI (high risk), 2) probable angina (intermediate risk), 3) low likelihood of angina (low risk), and then randomized to either receive MDCT immediately (MDCT group), or not (control). We compared diagnostic accuracy, length of stay in ER, admission rate, and major adverse cardiac events (MACE) and clinical diagnosis in 1 month after discharge from ED.

ELIGIBILITY:
Inclusion Criteria:

* Acute chest pain patient visiting emergency room

Exclusion Criteria:

* unstable vital sign
* renal failure
* ST elevation myocardial infarction
* uncontrolled arrhythmia
* hypersensitivity to contrast dye
* clinically no possibility of angina

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-04; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Admission rate
Unnecessary admission rate

SECONDARY OUTCOMES:
Stay time in emergency department
Diagnostic accuracy
MACE

CONTACTS AND LOCATIONS:
Overall Officials: Huk-Jae Chang, MD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang hospital, Sungnam-si, Kyungkido, South Korea